CLINICAL TRIAL: NCT04295863
Title: A Randomized Study Investigating the Pharmacokinetics of Standard Interval Dosing Compared to Extended Interval Dosing of Nivolumab or Pembrolizumab in Locally Advanced or Metastatic Cancers
Brief Title: Comparing Dosing Intervals of Nivolumab or Pembrolizumab in Locally Advanced or Metastatic Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-1718
Record Dates: First submitted 2020-02-14; First posted 2020-03-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- standard interval dosing (Experimental)
  Interventions: Drug: Nivolumab Standard; Drug: Pembrolizumab Standard
- extended interval dosing (Experimental)
  Interventions: Drug: Nivolumab Extended; Drug: Pembrolizumab Extended

INTERVENTIONS:
Drug: Nivolumab Standard — For patients on standard schedule dosing of nivolumab, therapy will consist of 240mg IV once every 2 weeks or 480mg IV once every 4 weeks
  Arms: standard interval dosing
Drug: Pembrolizumab Standard — For patients on standard schedule dosing of pembrolizumab, therapy will consist of 200mg IV once every 3 weeks or 400mg IV once every 6 weeks
  Arms: standard interval dosing
Drug: Nivolumab Extended — For patients on extended interval dosing of nivolumab therapy will consist of 240mg IV once every 4 weeks or 480mg IV once every 8 weeks
  Arms: extended interval dosing
Drug: Pembrolizumab Extended — For patients on extended interval dosing of pembrolizumab therapy will consist of 200mg IV once every 6 weeks
  Arms: extended interval dosing

SUMMARY:
A randomized research study of drugs nivolumab and pembrolizumab in patients with locally advanced or metastatic cancers. Based on data from earlier studies it appears that the drugs can be given less often then the currently approved schedule. This trial will compare drug levels from the blood from standard interval dosing levels versus taking the drugs less often.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advandced or metastatic cancer whose physician has determined they are candidates for treatment with nivolumab or pembrolizumab
* 18 years old or older
* Measurable disease per RECIST criteria

Exclusion Criteria:

* Patients who have previously received immune checkpoint inhibitors or investigational monoclonal antibody therapy.
* Patients whose treatment plan is to receive ipilimumab or other anti-CTLA4 monoclonal antibody in combination with either nivolumab or pembrolizumab.

  * Ipilimumab and nivolumab combination are not eligible for this trial.
  * (Note: Patients whose planned treatment is the combination of anti-PD-1 and tyrosine kinase inhibitor such as pembrolizumab-axitinib or the combination of traditional cytotoxic chemotherapy and anti-PD-1 are eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
Noninferiority margin of extended interval dosing compared to standard dosing | 2 years
  To assess the noninferiority of pharmacokinetic success, defined as drug trough levels above the target concentration of 1.5 µg/mL. Evaluable patients will be categorized as success or failure for this primary objective.

SECONDARY OUTCOMES:
Compare the efficacy of extended interval and standard interval dosing | 2 years
  To compare the correlation of extended interval and standard interval dosing, as based on a combination of time-to-treatment discontinuation (TTD) and overall survival (OS). This secondary analysis will include all patients who received at least one dose

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ratain, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois
  - SSM Health Cancer Care, Madison, Wisconsin